CLINICAL TRIAL: NCT04911673
Title: The Effect of Dark Chocolate and Music on Primary Dysmenorrhea
Brief Title: Effectiveness of Dark Chocolate and Music in Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, Ebru Baysal, Principal Investigator (Research Assistant), Celal Bayar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CelalBayar
Record Dates: First submitted 2021-05-20; First posted 2021-06-03 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Pain; Primary Dysmenorrhea; Menstrual Pain
Keywords: music; dark chocolate; dysmenorrhea; pain
MeSH Terms: conditions — Pain; Dysmenorrhea | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The name of students were listed in alphabetical order. The researchers gave each students a number. Then, the odd numbers were determined as the experimental and the even numbers as the control group with the lottery method. Using the table of random numbers, the intervention groups were divided into intervention group 1 (music therapy) and intervention group 2 (chocolate group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music group (Experimental): Participants listened a song with headphones that lasts 29 minutes and 32 seconds for four days (three days before menstruation and the first day of menstruation). The song was composed by Juan Martin Saavedra.
  In the first month, music group was filled the State Anxiety Inventory (SAI) between 10 and 20th of the menstruation that SAI consists of 20 statements that ask people to describe how they generally feel. In the second month, pain scores were measured on the first day of menstruation using a visual analogue scale (VAS) of 10 cm (0 no pain at all, and 10 the worst possible pain) and Trait Anxiety Inventory (TAI) was filled to assess the anxiety.In the third month, after the participants were listening the music in three days before menstruation and the first day of menstruation (during four days), pain scores were measured on the first day of menstruation using VAS and TAI was filled to assess the anxiety.
  Interventions: Behavioral: music
- Chocolate group (Experimental): Participants ate 40 mg of dark chocolate with 60% cocoa per day for four days (three days before menstruation and the first day of menstruation) that was given by researchers to them. In the first month, chocolate group was filled the SAI to assess state anxiety between 10 and 20th of the menstruation.In the second month, pain scores were measured on the first day of menstruation using VAS and TAI was filled to assess the trait anxiety.In the third month, after the participants were eating 40 mg of dark chocolate per day in three days before menstruation and the first day of menstruation (during four days/total 160 mg), pain scores were measured on the first day of menstruation using VAS and TAI was filled to assess the anxiety.
  Interventions: Dietary Supplement: Chocolate group
- Control group (No Intervention): Control group had no intervention. In the first month, control group was filled the SAI to assess state anxiety between 10 and 20th of the menstruation. In the second month, pain scores were measured on the first day of menstruation using VAS and TAI was filled to assess the trait anxiety. In the third month, pain scores were measured on the first day of menstruation using VAS and TAI was filled to assess the anxiety.

INTERVENTIONS:
Behavioral: music — Participants listened a song with headphones that lasts 29 minutes and 32 seconds for four days (three days before menstruation and the first day of menstruation).
  Arms: Music group
Dietary Supplement: Chocolate group — Participants ate 40 mg of dark chocolate with 60% cocoa per a day for four days (three days before menstruation and the first day of menstruation) that was given by researchers to them.
  Arms: Chocolate group

SUMMARY:
Primary dysmenorrhea (PD) is a pain that occurs in the menstrual period without pathological pelvic disorder. Excessive prostaglandin release causes uterine contraction and leads to uterine hypoxia and ischemia, which results in extreme abdominal cramps and pain. Music therapy is one of the complementary treatment methods in the management of pain for PD which is an intervention that is not expensive and has no side effects. Another complementary treatment method is for PD is chocolate. In the literature; there have a few studies about the effect of the music and dark chocolate on the primary dysmenorrhea but no studies have been conducted to evaluate the effects of the music and dark chocolate on PD.

The following is the protocol for a randomized controlled clinical trial, where an experimental group 1 listened to a 30-minute song, an experimental group 2 ate dark chocolate and a control group had no intervention for the same time and conditions. The aim of this study is to determine the effect of dark chocolate and music on PD. This pain measured through a 10 cm Visual Analogue Scale (VAS) in nursing students from the Faculty of Health Sciences at the Manisa Celal Bayar University, Manisa, Turkey. Additionally, State-Trait Anxiety Inventory (STAI) was used to assess the trait and state anxiety.

DETAILED DESCRIPTION:
Primary Dysmenorrhea (PD) is defined as cramping pain in the lower abdomen, which occurs before or during menstruation without pelvic diseases. Contraceptive pills and non steroidal anti inflammatory drugs are commonly used in the treatment of PD. International (66.5% to 92.5%) and Turkey (87.7% to 80.1%) in the studies among university students show that a high percentage of dysmenorrhea. Dysmenorrhea negatively affects the school absenteeism of girls, their academic success and causes a lack of concentration. The rate of using pain medication due to dysmenorrhea is high among students. Music therapy has been shown to be effective in relaxing the mind and body, relieving anxiety, enhancing security, and increasing pain thresholds. Dark chocolate contains copper, which is used by the body to synthesize neurotransmitters called collagen and endorphins. Endorphin hormone is an analgesic and natural sedative to reduce pain intensity such as menstrual pain.

This randomized clinical trial was designed to determine the effect of eating dark chocolate and listening music on PD, compared to a control group that no intervention in women of 18 years or older from the the Faculty of Health Sciences at the Manisa Celal Bayar University, Manisa, Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Legal and cognitive capacity for informed consent.
* Suffering from primary dysmenorrhea (low abdominal pain associated to menses). (five and above in VAS)
* Being able to understand and use the measuring tools and questionnaires.
* 18-25 years old
* Studying in Manisa Celal Bayar University, Faculty of Health Sciences, Department of Nursing, in the 2020-2021 academic year, in the 1st, 2nd, 3rd and 4th grades,

Exclusion Criteria:

* Previous diagnosis of pelvic pathology.
* Diagnosis of hearing impairment.
* Diagnosis of neurologic or endocrinological disease.
* Psychiatric condition diagnosed.
* Known or reported previous substance abuse.
* Current use of psychiatric drugs.
* Cancer diagnosis
* Diagnosed chronic diseases such as diabetes mellitus or heart disease.
* Previous advance musical training (defined as any form of music training in addition to that received during normal school classes).
* Irregular menstrual cycles.
* Previous pregnancy.
* Current use of any hormonal contraceptive therapy
* Having allergy to chocolate
* Being obese
* Taking vitamin supplements
* Students who do not agree to participate in the research

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 18-25 years old
Enrollment: 84 (Actual)
Dates: Start 2021-01-30 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Description of the students' demographics and clinical backgrounds. | It was implemented on the first day of the study and it took approximately 10-15 minutes to fill out the form.
  Questions about the sociodemographic characteristics and dysmenorrhea characteristics of the students were asked using the individual identification form developed by the researchers in line with the literature.
To evaluate pain severity secondary to dysmenorrhea in the first day of menstruation through a Visual Analogue Scale (VAS). | The first day of the menstrual cycle 1 (each cycle is 28 days) and it is the baseline data.
  We asked them to determine the severest pain score they felt on the first day of menstruation according to the VAS scale. The highest pain score that can be obtained on the VAS scale is 10 and the lowest is 0.
To evaluate the effect of dark chocolate consumption in reducing the pain severity secondary to dysmenorrhea in the first day of menstruation through a Visual Analogue Scale (VAS). | The first day of the menstrual cycle 2 (each cycle is 28 days) and it is the post intervention data.
  We asked them to eat dark chocolate and determine the severest pain score they felt on the first day of menstruation according to the VAS scale. The highest pain score that can be obtained on the VAS scale is 10 and the lowest is 0. Participants ate 40 mg of dark chocolate per day for four days (three days before menstruation and the first day of menstruation) that was given by researchers to them.
To evaluate the effect of music consumption in reducing the pain severity secondary to dysmenorrhea in the first day of menstruation through a Visual Analogue Scale (VAS). | The first day of the menstrual cycle 2 (each cycle is 28 days) and it is the post intervention data.
  We asked them listen to music and to determine the severest pain score they felt on the first day of menstruation according to the VAS scale. The highest pain score that can be obtained on the VAS scale is 10 and the lowest is 0. Students listened a song with headphones that lasts 29 minutes and 32 seconds for four days (three days before menstruation and the first day of menstruation). Participants were instructed to avoid using cellphones or other activities during the time of the intervention.
To evaluate anxiety level in the first day of first menstruation cycle through State Anxiety Inventory (SAI). | The first day of the menstrual cycle 1 (each cycle is 28 days) and it is the baseline data.
  In the first day of first menstrual cycle, students was filled the State Anxiety Inventory (SAI) that SAI consists of 20 statements that ask people to describe how they generally feel. Each question is rated on a 4-point scale (not at all, somewhat, moderately so, very much so). The SAI varies from a minimum score of 20 to a maximum score of 80. SAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).
To evaluate the effect of dark chocolate consumption in reducing the anxiety level of students with dysmenorrhea using State-Trait Anxiety Inventory (STAI). | The first day of the menstrual cycle 2 (each cycle is 28 days) and it is the post intervention data.
  We asked them to eat dark chocolate and filled the State Anxiety Inventory (SAI)in the first day of first menstrual cycle. The SAI consists of 20 statements that ask people to describe how they generally feel. Each question is rated on a 4-point scale (not at all, somewhat, moderately so, very much so). The SAI varies from a minimum score of 20 to a maximum score of 80. SAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).
To evaluate the effect of the music in reducing the anxiety level of students with dysmenorrhea using State-Trait Anxiety Inventory (STAI). | The first day of the menstrual cycle 2 (each cycle is 28 days) and it is the post intervention data.
  We asked them to listen the music and filled the State Anxiety Inventory (SAI)in the first day of first menstrual cycle. The SAI consists of 20 statements that ask people to describe how they generally feel. Each question is rated on a 4-point scale (not at all, somewhat, moderately so, very much so). The SAI varies from a minimum score of 20 to a maximum score of 80. SAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).

CONTACTS AND LOCATIONS:
Overall Officials: EBRU BAYSAL, PhD, Principal Investigator — Manisa Celal Bayar University
Locations (1):
- Ebru Baysal, Manisa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No